CLINICAL TRIAL: NCT03655938
Title: Piezocision-assisted Orthodontic Treatment Combined With Alveolar Bone Regeneration : a Prospective Study
Brief Title: Piezocision-assisted Orthodontic Treatment Combined With Alveolar Bone Regeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P2016-1 In-OP WP2
Record Dates: First submitted 2018-06-11; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Patients Requiring Mandible Orthodontic Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Piezocision combined minimally invasive alveolar bone regeneration — The piezocision surgery was performed two weeks after orthodontic appliance placement. The patients received local anesthesia in mandibular arch and vertical interproximal incisions were made below the interdental papillae in the midline, from the mesial aspect of each canine and in between each of the posterior lower teeth. The periostium was then released in order to create two subperiotal envelopes connecting the vertical incisions together. Thereafter, corticotomies were performed in the region of the incisions with a piezotome (Acteon, Merignac, France) and the envelopes were filled with a beta tricalcium phosphate, a resorbable biomaterial in order to thicken the buccal bone plate. Resorbable 5-0 sutures were used to close the flaps. Careful tooth brushing and the use of a mouthwash (chlorhexidine 0.2% Perio-Aid, Dentaid Benelux, Houten, Netherlands) were recommended for 7 days.

SUMMARY:
This study was designed to enroll a series of 10 consecutive patients who met the inclusion criteria. Patients were treated in the Department of Orthodontics and Dento-Facial Orthodopedics of the University of Liège. Two senior's orthodontists and two senior's periodontists were involved in the orthodontic treatment and in the surgical procedures respectively. All clinical, radiographic and periodontal measurements and all orthodontic parameters were performed at baseline and after the orthodontic treatments. Tree examiners collected the overall data.

ELIGIBILITY:
Inclusion criteria:

* Patients requiring at least mandible orthodontic treatment (both arches)
* Patient presenting alveolar bone thickness < XX mm
* Adult patients with completed growth based on the Cervical Vertebral Maturation Method (CVM) as described by Baccetti et al. (Baccetti et al. 2002)
* Minimal to moderate mandibular anterior crowding at baseline (irregularity index≤6) (Little 1975)
* American Society of Anesthesiology I or II (I = Normal healthy patient; II = Patients with mild systemic disease)
* Adequate dento-oral health (i.e., the absence of periodontal diseases, peri-apical infection, or untreated caries).

Exclusion criteria were as follows:

* Controlled periodontitis with a loss of alveolar support > 10%
* Gingival recession > 2 mm
* Smokers
* Altered bone metabolism (e.g., due to anti-resorptive drug, steroid or immunosuppressant use)
* Mental or motor disabilities
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Radiographic change from Baseline and after 1year | Baseline and after 1year
  The patients underwent baseline and post treatment CBCT scans (Somaton® Emotion; Siemens, Munich, Germany). Measurements of the alveolar bone changes in the lower front region on pre- and post- treatment CT volumes were done by reformatting the orthogonal slices, along the sagittal, coronal and axial length axes of each individual tooth. A strict vestibular bone level measurement (sagittal slice) and three alveolar bone width measurements at crestal level, 3mm from the crest and 6mm from the crest (axial slices) were performed per individual tooth. In addition, CT images were analyzed in using a dedicated platform in an image processing software (MeVisLab, MeVis Medical Solutions AG, Bremen,Germany) where pre- and post-treatment volumes were superposed using rigid image registration. Semi-automatically segmentation using region growing with same seed-point and threshold value for both scans, was followed with a hole-filling algorithm to obtain segmented volumes of the cropped image in

SECONDARY OUTCOMES:
Periodontal Evaluation | Baseline and after 1 year
  The following clinical parameters were measured at baseline and after the orthodontic treatments: recession depths (RDs), pocket depth, plaque index (PI) and papilla bleeding index (PBI). A recession score was calculated by summing the recession depths. Next, the presence of gingival scars due to the overall treatment of each patient was categorized as an absence of scars, point-shape scars or linear-shape scars. Full periodontal charting (probing in four sites per tooth) was performed in all patients before and after the treatment; the results were expressed as score per sextant.
Patient assessment | Baseline and after 1year
  The patient-centered outcomes were recorded using a Visual Analog Scale questionnaire that employed a 0-10 graduated scale. The following parameters were collected: apprehension before treatment (scale ranges, minimum=0 and maximum=10) scores), pain level after treatment and daily analgesic consumption following orthodontic appliance placement and piezocision (scale ranges, minimum=0 and maximum=10). After the overall treatment, the levels of satisfaction in terms of the final result (scale ranges, minimum=0 and maximum=10), the treatment duration and whether the patient would recommend the procedure to a friend were assessed (scale ranges, Yes=0 and No=10). Finally, the patients were asked whether they would undergo the treatment again (scale ranges, Yes=0 and No=10).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU University of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charavet C, Lecloux G, Vandenberghe B, Lambert F. Buccal bone regeneration combined with piezocision in adult orthodontic patients: Clinical, 3D radiographic, and patient-reported outcomes. J Stomatol Oral Maxillofac Surg. 2021 Dec;122(6):549-556. doi: 10.1016/j.jormas.2020.10.005. Epub 2020 Oct 22. PMID 33289660